CLINICAL TRIAL: NCT02766517
Title: LY2951742 Biomarker Study in Patients With Migraine
Brief Title: Biomarker Study in Participants With Migraine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16235; I5Q-MC-S001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2017-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capsaicin (Experimental): Single topical dose of capsaicin
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin — Administered topically

SUMMARY:
This is a study of participants with a diagnosis of migraine who completed another clinical trial NCT02163993. The participants received either LY2951742 or placebo. This study NCT02766517 will evaluate how certain biomarkers may be related to the participant's response in study NCT02163993. The study will last about five days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with migraine who have previously participated in study NTC02163993 and received one of the selected doses of galcanezumab or placebo
* Have suitable skin characteristics for the dermal capsaicin challenge

Exclusion Criteria:

* Have a history of significant allergies, in particular to ethanol or sensitivity to the fruits of capsicum plants (for example, chili peppers)
* Have eczema, scleroderma, psoriasis, dermatitis, keloids, tumors, ulcers, burns, flaps, or grafts on their forearm or other abnormality of the skin which may interfere with the study assessments
* Cannot avoid excess tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and cannot cover forearms for 24 hours prior to each treatment period
* Have excessive hair growth on the volar surface of the forearm or participants currently using lotions, oils, depilatory preparations, or other topical treatments on a regular basis which cannot be discontinued for the duration of the study; has used any topical treatments within 7 days of the start of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - Arizona Research Center, Phoenix, Arizona
  - Pharmacology Research Institute, Newport Beach, Encino, California
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - Pharmacology Research Institute, Newport Beach, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, Newport Beach, California
  - Medical Center for Clinical Research, San Diego, California
  - California Clinical Trials, San Diego, California
  - Avail Clinical Research LLC, DeLand, Florida
  - Psychiatric Inst of Florida-Clinical Neuroscience Solutions, Orlando, Florida
  - PharmaSite Research Inc, Baltimore, Maryland
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland
  - Rochester Clinical Research, Inc., Rochester, New York
  - CNS Health Care, Memphis, Tennessee
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with migraine who had previously participated in the Phase 2 galcanezumab study, NCT02163993 [I5Q-MC-CGAB], and received either 120 milligram (mg) or 300 mg galcanezumab or placebo, with suitable skin characteristics for the dermal capsaicin challenge, were included in the I5Q-MC-S001 (NCT02766517) trial.
Groups:
- Placebo: Participants who received placebo in previous study I5Q-MC-CGAB administered with 1000 microgram (mcg) capsaicin solution and vehicle topically in current study.
- 120 mg Galcanezumab: Participants who received 120 mg galcanezumab (LY2951742) in previous study I5Q-MC-CGAB administered with 1000 mcg capsaicin solution and vehicle topically in current study.
- 300 mg Galcanezumab: Participants who received 300 mg galcanezumab (LY2951742) in previous study I5Q-MC-CGAB administered with 1000 mcg capsaicin solution and vehicle topically in current study.
Period: Overall Study
Arm/Group | Placebo | 120 mg Galcanezumab | 300 mg Galcanezumab
Started | 19 | 9 | 9
Completed | 19 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants who received placebo in previous study I5Q-MC-CGAB administered with 1000 mcg capsaicin solution and vehicle topically in current study.
- Total: Total of all reporting groups
Arm/Group | Placebo | 120 mg Galcanezumab | 300 mg Galcanezumab | Total
Number analyzed (Participants) | 19 | 9 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (13.0) | 47.6 (7.8) | 42.3 (15.0) | 43.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 7 | 28
  Male | 4 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6
  Not Hispanic or Latino | 16 | 9 | 6 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 4 | 13
  White | 13 | 4 | 5 | 22
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 9 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Capsaicin-Induced Dermal Blood Flow (DBF)
Description: Change from pre-capsaicin DBF adjusting for vehicle at 30 minutes is reported. The capsaicin induced dermal blood flow (DBF) was measured by laser Doppler imaging (LDI).
Time Frame: Baseline (pre-capsaicin) and on assessment day over approximately one hour, after at least a 4 month wash out from treatment in study NCT02163993
Population: All enrolled participants who have evaluable pharmacodynamics data.
Measure: Mean (Standard Deviation); unit: Flux mean
Arm/Group | Placebo | 120 mg Galcanezumab | 300 mg Galcanezumab
Number analyzed (Participants) | 19 | 7 | 9
Flux mean | 606.1 (615.6) | 599.5 (514.7) | 689.2 (552.3)

2. Primary Outcome: Plasma Calcitonin Gene-Related Peptide (CGRP) Levels
Description: The mean Plasma Calcitonin Gene-Related Peptide levels were reported.
Time Frame: On assessment day over approximately one hour, after at least a 4 month wash out from treatment in study NCT02163993
Population: All enrolled participants who have evaluable pharmacodynamics data.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | 120 mg Galcanezumab | 300 mg Galcanezumab
Number analyzed (Participants) | 19 | 9 | 9
picogram per milliliter (pg/mL) | 1.748 (1.322) | 1.082 (0.261) | 1.370 (0.318)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 3
Arm/Group | Placebo | 120 mg Galcanezumab | 300 mg Galcanezumab
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/19 | 1/9 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | 120 mg Galcanezumab (N=9) | 300 mg Galcanezumab (N=9)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 2 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.